CLINICAL TRIAL: NCT01625715
Title: A Prospective, Randomized, Case Controlled, Pilot Study to Evaluate the Effect of Ketotifen on the Adverse Events Associated With Peanut Desensitization in Children With Peanut Allergies.
Brief Title: Pilot Study to Evaluate the Effect of Ketotifen on the Adverse Events Associated With Peanut Desensitization
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gordon Sussman Clinical Research (Other)
Collaborators: Mast Cell Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCP-001
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Peanut Allergies in Children
Keywords: peanut allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Ketotifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case control (No Intervention): Routine therapy during peanut desensitization
- ketotifen (Experimental): rising doses of ketotifen
  Interventions: Drug: Ketotifen

INTERVENTIONS:
Drug: Ketotifen — titrated dose: 1 mg once a day, then 1 mg twice a day then 2 mg twice a day
  Arms: ketotifen

SUMMARY:
The primary objective of this study is to evaluate, compared to non-treatment, the impact of a titrated dose (1 mg once a day, then 1 mg twice a day and finally a full 2 mg twice a day) of ketotifen on the adverse event profile emerging from a rapid peanut desensitization protocol, in children with established peanut allergy.

DETAILED DESCRIPTION:
The development of a safe oral peanut challenge procedure permits patients that do not have severe life threatening allergic reactions, to be safely desensitized with the ability to maintain peanut tolerance . The peanut desensitization procedure is however associated with unpleasant allergic side effects mainly gastrointestinal and cutaneous manifestations. The use of premedication drugs may lessen these side effects and facilitate the peanut desensitization procedure. Ketotifen is a fast acting, noncompetitive, H1-receptor blocker (antihistamine/inverse agonist) that also inhibits the release of mediators from mast cells involved in hypersensitivity reactions.

The study will enroll 6 (4 in the peanut treatment group, 2 in the control group) children with a known history of peanut allergies. The treated subjects will be randomized in a 2:1 ratio into either a pre-treatment group (final dose of 2 mg bid ketotifen) or a control group. All subjects will undergo a one-day peanut desensitization protocol designed to enable the subject to tolerate 50 mg of peanut flour (initial escalation phase). After the initial escalation day achieving up to 50 mg of peanut flour, the dosing build-up will occur every two weeks through 44 weeks. Subjects will ingest the 50mg and increased doses of peanut flour at home (every day for 2 weeks) between each dose escalation. The target dose is 8000 mg of peanut flour. A maintenance dose will be given for 4 weeks following the last (highest dose) visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years, all of either sex, any race, any ethnicity at the time of the initial visit
* The presence of IgE specific to peanuts (a positive skin prick test to peanuts (diameter of wheal >3.0 mm) and a positive in vitro IgE [CAP-FEIA] > 7 kUA/L
* A history of significant clinical symptoms occurring within 60 minutes after ingesting peanuts
* Provide signed informed consent.

Exclusion Criteria:

1. History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise (Cyanosis or SpO2 < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence)
2. Currently participating in a study using an investigational new drug
3. Participation in any interventional study for the treatment of food allergy in the past 12 months
4. Subjects with a known oat or wheat (because of potential cross contamination with oat) food allergy will be excluded
5. Poor control or persistent activation of atopic dermatitis
6. Moderate to severe persistent asthma
7. Currently being treated with greater than medium daily doses of inhaled corticosteroids, as defined by the NHLBI guidelines
8. Inability to discontinue antihistamines for skin testing
9. History of epilepsy or seizures
10. Diabetes

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Event leading to discontinuation | up to 12 months
  Treatment with peanut flour causes ADRs that lead to treatment discontinuation.

SECONDARY OUTCOMES:
Clinical Global Assessment | 12 months
  Investigator's assessment of treatment impact on moderating adverse reactions associated with desensitization.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon L Sussman, MD, Principal Investigator
Locations (1):
- GSCRI, Toronto, Ontario, Canada